CLINICAL TRIAL: NCT00214279
Title: MMF Monotherapy and Immune Regulation in Kidney Transplant Recipients: Part 1 Steroid Withdrawal
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2002-040; CEL340
Record Dates: First submitted 2005-09-14; First posted 2005-09-21 (Estimated); Last update posted 2012-06-26 (Estimated); Status verified 2012-06

CONDITIONS: Renal Transplantation

ARMS (2):
- 1 (No Intervention): Remain on 3-drug standard of care immunosuppression including prednisone
- 2 (Experimental): Corticosteroid withdrawal / prednisone taper over 14 weeks
  Interventions: Drug: Corticosteroid withdrawal

INTERVENTIONS:
Drug: Corticosteroid withdrawal — prednisone withdrawal, with maintenance mycophenolate mofetil therapy and either cyclosporine or tacrolimus
  Arms: 2

SUMMARY:
Part 1 of the study is to gradually withdraw steroids in a group of 50 older renal transplant recipients, converting then from the 3 drug regimen to a 2 drug regimen (cyclosporine and MMF), while carefully monitoring their graft function. 25 subjects would serve as control patients in the study and would remain on the 3 drug regimen (steroids, cyclosporine and MMF). Immunologic status will be determined before and after IS withdrawal using a delayed-type hypersensitivity (DTH) transfer test previously described in the original submission. Both the steroid withdrawal subjects and the control subjects will undergo the DTH testing throughout the 3 years of study participation.

ELIGIBILITY:
Inclusion Criteria:

* Patient who have received a kidney transplant during the "MMF era"
* Patients who have stable graft function indicated by a serum creatinine of < 1.8 mg/dl, or a calculated creatinine clearance of > 50 ml/minute

Exclusion Criteria:

* Patients who have had > 1 rejection episode,
* Patients who have had a rejection episode within the past year;
* Patients who are steroid dependent due to pre-existing disease (for example, RA or SLE

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2002-05; Primary Completion 2007-11 (Actual); Study Completion 2007-11 (Actual)

PRIMARY OUTCOMES:
Incidence of Allograft rejection | 3 years

SECONDARY OUTCOMES:
Renal function as determined by serum creatinine | measure after 36 months
Allograft Survival | 3 years
Immunological function as determined by Trans-vivo delayed hypersensitivity assay (TV-DTH) | Day 0 (pre-transplant)
  Research assay done to determine correlation between the status of donor specific regulation (DSR) and rates of rejection in both arms of the study.

CONTACTS AND LOCATIONS:
Overall Officials: Hans Sollinger, MD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- Unversity of Wisconsin, Madison, Wisconsin, United States